CLINICAL TRIAL: NCT02933502
Title: An Open-label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment With DSXS 1538b Topical Product Applied Once-daily in Patients With Moderate to Severe Scalp Psoriasis
Brief Title: Safety Study in Patients With Scalp Psoriasis Suppression Following Maximal Use Treatment With Topical Product
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1538b
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSXS topical product (Experimental): treatment with DSXS once daily for 28 days
  Interventions: Drug: DSXS topical product

INTERVENTIONS:
Drug: DSXS topical product — treatment daily for 28 days
  Other Names: Active

SUMMARY:
An Open-Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use DSXS topical product (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Moderate to SevereScalp Psoriasis

DETAILED DESCRIPTION:
* Evaluate the potential of DSXS topical product to suppress HPA axis function in patients with moderate to severe scalp psoriasis.
* Evaluate the efficacy parameters and adverse event (AE) profiles of DSXS topical product administered to patients with moderate to severe scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 12-17 years of age.

Exclusion Criteria:

* Females who are pregnant, nursing, planning to become pregnant during the duration of the study, or if of child-bearing potential and sexually active and not prepared to use appropriate contraceptive methods to avoid pregnancy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSXS Topical Product
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DSXS Topical Product
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Percent Scalp Affected with Plaque Psoriasis [Mean (Standard Deviation); unit: percent of scalp] | 28.3 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to stimulation
Time Frame: day 28
Population: Two patients who had normal adrenal function at baseline, used at least 21 doses of the study product, and had data from a post-treatment cortisol response test were included in the analysis. One patient was excluded from the analysis of HPA axis suppression owing to abnormal adrenal function at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical Product
Number analyzed (Participants) | 2
Participants
  Yes | 0
  No | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DSXS Topical Product
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT02933502/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT02933502/SAP_001.pdf